CLINICAL TRIAL: NCT05771194
Title: Analysis of Postoperative Ocular Surface Changes and Intervention Effect After PPV in MGD Dry Eye Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Bojie Hu, Director,head of ophthalmology;Principal Investigator, Tianjin Medical University Eye Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hbj112233
Record Dates: First submitted 2023-02-19; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Meibomian Gland Dysfunction of Unspecified Eye, Unspecified Eyelid
Keywords: Meibomian gland dysfunction; Dry eye; Non-invasive ocular surface analyser; Pars plana vitrectomy; ,Meibomian gland massage
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Group A received conventional preoperative and postoperative anti-infective therapy.
  Interventions: Drug: Routine preoperative and postoperative anti-infection therapy
- group B (Active Comparator): On the basis of group A,Group B was given 0.1% sodium hyaluronate eye drops 4 times daily for 3 days before surgery (Jiang Xi, Zhen Shiming Pharmaceutical Co., Ltd.) and 3 months after surgery, and one cleaning, hot compresses and massage of the meibomian gland.
  Interventions: Drug: Routine preoperative and postoperative anti-infection therapy; Drug: artificial tear therapy; Procedure: Cleaning, hot compresses and massage of the meibomian gland

INTERVENTIONS:
Drug: Routine preoperative and postoperative anti-infection therapy — received gatifloxacin eye drops (Otsuka Pharmaceutical Co., Ltd.) 4 times daily and gatifloxacin eye ointment once every night (Shenyang Xing Qi Pharmaceutical Co., Ltd) for 3 days before surgery. Postoperatively, gatifloxacin eye drops were administered 4 times daily, 0.1% fluorometholone (San Tian Pharmaceutical Co., Ltd., China) was administered 4 times daily, and pranoprofen (Qian Su Pharmaceutical Co., Ltd., Japan) was administered 4 times daily. The doses of the above three drugs were reduced each week. The compound tropicamide was administered once a day (Shentian Pharmaceutical Co., Ltd., China). All of the above procedures were stopped 1 month after surgery.
Drug: artificial tear therapy — given 0.1% sodium hyaluronate eye drops 4 times daily for 3 days before surgery (Jiang Xi, Zhen Shiming Pharmaceutical Co., Ltd.) and 3 months after surgery.
  Arms: group B
Procedure: Cleaning, hot compresses and massage of the meibomian gland — Group B used a steam eye mask (Your Ga Run Fang, Shang Hai Run Mu Industrial Co., Ltd.) for 20 minutes 3 days before surgery. Sterile cotton swabs were used to apply physiological saline to the eyelid for local cleaning, and the secretions and phosphorus debris on the surface of the eyelid margin were removed to fully expose the meibomian gland. Meibomian gland tweezers were used to squeeze from the root of the gland toward the opening to expel the secretions; each gland was expressed twice. After the operation, an appropriate amount of gatifloxacin cream (Shen Yang Xing Qi Pharmaceutical Co., Ltd.) was applied to the conjunctival sac to prevent infection. Hot towels (40°C) were applied to the eyes for 10 minutes every morning and evening for 3 days before the operation.
  Arms: group B

SUMMARY:
AIM: To observe ocular surface changes after phacovitrectomy in patients with mild to moderate meibomian gland dysfunction (MGD)-type dry eye and track clinical treatment response using a Keratograph 5M and a LipiView interferometer.

METHODS: Forty cases were randomized into control group A and treatment group B; the latter received meibomian gland treatment 3 days before phacovitrectomy and sodium hyaluronate before and after surgery. The average non-invasive tear film break-up time (NITBUTav), first non-invasive tear film break-up time (NITBUTf), non-invasive measured tear meniscus height (NTMH), meibomian gland loss (MGL), lipid layer thickness (LLT) and partial blink rate (PBR) were measured preoperatively and 1 week, 1 month and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dry eye
* Clinical diagnosis for MGD

Exclusion Criteria:

* eye trauma or eye surgery within the prior 6 months
* use of drugs that affect tear secretion and the stability of the tear film (including anti-glaucoma drugs, cortisol drugs, etc.) within the prior 6 months
* other diseases that affect the function of the eye surface, such as meibomian gland cysts, blepharitis, eyelid valgus, incomplete closure, chronic tear cystitis, corneal disease, glaucoma, or optic neuropathy
* intraoperative suture fixation or closure of a corneal, conjunctival, or scleral incision
* long-term postoperative intraocular hypertension that could not be controlled easily with oral drugs and required puncture and drainage through the anterior chamber
* postoperative corneal epithelial defects lasting more than 1 week or necessitating the use of contact lenses for treatment
* the need for a second operation during the study follow-up eye trauma or eye surgery within the prior 6 months
* use of drugs that affect tear secretion and the stability of the tear film (including anti-glaucoma drugs, cortisol drugs, etc.) within the prior 6 months
* other diseases that affect the function of the eye surface, such as meibomian gland cysts, blepharitis, eyelid valgus, incomplete closure, chronic tear cystitis, corneal disease, glaucoma, or optic neuropathy
* intraoperative suture fixation or closure of a corneal, conjunctival, or scleral incision
* long-term postoperative intraocular hypertension that could not be controlled easily with oral drugs and required puncture and drainage through the anterior chamber
* postoperative corneal epithelial defects lasting more than 1 week or necessitating the use of contact lenses for treatment
* the need for a second operation during the study follow-up

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
The average non-invasive tear film break-up time | 5minutes to 10 minutes
  The NITBUT values were measured using a non-invasive ophthalmic analyser; the patients were instructed to blink 2 times after a normal blink, focus their eyes, and then refrain from blinking until the Placido ring projected onto the cornea was broken; the duration was recorded.

SECONDARY OUTCOMES:
lipid layer thickness | 1minutes to 5 minutes
  The LipiView interferometer was used for examination under natural light. The patient was in a sitting position, and the mandible and forehead were against the jaw bracket and the forehead bracket, respectively. The aiming frame was aligned between the pupil and the lower eyelid margin; the position was adjusted until the reflection of the lower eyelashes was clear. Patients were asked to gaze at the light source for approximately 20 s and blink normally. The average LLT were recorded.
non-invasive measured tear meniscus height | 1minutes to 5 minutes
  The lacrimal river was imaged, and the height of the lacrimal river directly below the centre of the pupil was measured with the built-in measurement tool of the system. Each patient was examined by the same ophthalmologist three times, and the average of the three measurements was used as the final result.
meibomian gland loss | 1minutes to 5 minutes
  The Meibo-Scan mode was selected. Then, the upper and lower eyelids were turned outward, and morphological images of the meibomian glands were obtained under an infrared light source. The shortening and loss of meibomian glands were observed and recorded on the following scale: The absence of meibomian gland loss (MGL) corresponded to a score of 0 point, an MGL ratio of less than 1/3 was assigned 1 point, an MGL ratio of 1/3 to 2/3 received 2 points, and a ratio of >2/3 received 3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Jie Hu, Study Chair — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No